CLINICAL TRIAL: NCT00433927
Title: Multicenter Randomized Trial Evaluating FOLFIRI Plus Cetuximab Versus FOLFIRI Plus Bevacizumab in First Line Treatment of Metastatic Colorectal Cancer.
Brief Title: 5-FU, Folinic Acid and Irinotecan (FOLFIRI) Plus Cetuximab Versus FOLFIRI Plus Bevacizumab in First Line Treatment Colorectal Cancer (CRC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PD Dr. med. Volker Heinemann (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor-Investigator, PD Dr. med. Volker Heinemann, Sponsor Delegated Person, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIRE-3
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Neoplasm Metastasis; Colorectal Cancer
Keywords: metastatic
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; Cetuximab; Bevacizumab

ARMS (2):
- Arm A (Active Comparator): FOLFIRI plus Cetuximab
  Interventions: Drug: 5-FU; Drug: folinic acid; Drug: irinotecan; Drug: cetuximab
- Arm B (Active Comparator): FOLFIRI plus Bevacizumab
  Interventions: Drug: 5-FU; Drug: folinic acid; Drug: irinotecan; Drug: bevacizumab

INTERVENTIONS:
Drug: 5-FU — 5-FU 400 mg/m² Bolus day 1 5-FU 2400 mg/m² iv over 46 h day 1-2
Drug: folinic acid — Folinsäure (racemisch) 400 mg/m² iv, 120 min d 1
Drug: irinotecan — Irinotecan 180 mg/m² iv, 30 - 90 min day 1
Drug: cetuximab — Cetuximab initial 400mg/m² as 120 min infusion, than 250 mg/m² iv as 60 min infusion d 1 + 8
  Arms: Arm A
Drug: bevacizumab — Bevacizumab 5 mg/kg iv over 30 to 90 minutes d 1
  Arms: Arm B

SUMMARY:
The FIRE-3 trial is a multicenter randomized phase III trial investigating 5-FU, folinic acid and irinotecan (FOLFIRI) plus cetuximab versus FOLFIRI plus bevacizumab in first line treatment of metastatic colorectal cancer. Planned accrual is 284 evaluable patients per treatment arm. The primary study endpoint is objective response rate. Secondary endpoints are median progression free survival, median overall survival, safety, and secondary resection rate.

ELIGIBILITY:
Inclusion Criteria:

* KRAS-Wildtype status
* Histologically confirmed adenocarcinoma of the colon or rectum.
* Stage IV disease.
* ECOG 0-2.
* Patients considered suitable for application of chemotherapy.
* Age 18 - 75 years.
* In- or outpatient treatment.
* Estimated life expectancy > 3 months.
* Measurable index lesion according to RECIST criteria. Evaluation of tumor manifestations ≤ 2 weeks prior to treatment start.
* Effective contraception.
* Adequate hematologic function: leukocytes >= 3000/µl, neutrophils >= 1500/µl, platelets >= 100.000/µ, and hemoglobin >= 9g/dl.
* Bilirubin <= 1,5x upper limit of normal (ULN).
* ALAT and ASAT <= 2,5x ULN, in case of liver metastases <= 5x ULN.
* Serum creatinine <= 1,5x ULN.
* No operations within 4 weeks prior to treatment start. No cytologic biopsies within 1 week prior to treatment start. Operation sequels need to be completely healed. Major operations must not be expected at time of study begin, except for potential secondary resection of liver metastases. In case of secondary resection of liver metastases, bevacizumab must be discontinued 6-8 weeks prior to surgery.
* No relevant toxicities due to prior medical treatment at time of study entry.

Exclusion Criteria:

* KRAS-Mutation of the tumor
* Prior treatment directed against the epidermal growth factor receptor (EGFR).
* Prior treatment with bevacizumab.
* Prior chemotherapy for colorectal cancer, except for adjuvant chemotherapy dating back > 6 months prior to study entry.
* Experimental medical treatment within 30 days prior to study entry.
* Known hypersensitivity reaction to any study medication.
* Pregnant or breast feeding women (pregnancy needs to be excluded by testing of beta-HCG).
* Known or suspected cerebral metastases.
* Clinically significant coronary heart disease, myocardial infarction within the last 12 months or high risk of uncontrolled arrhythmia.
* Acute or subacute ileus, chronic inflammatory bowel disease or chronic diarrhea.
* Symptomatic peritoneal carcinosis.
* Severe chronic wounds, ulcera or bone fracture.
* Uncontrolled hypertension.
* Severe proteinuria (nephrotic syndrome).
* Arterial thromboembolic events or hemorrhage within 6 months prior to study entry (except tumor bleeding surgically treated by tumor resection).
* Bleeding diatheses or coagulopathy.
* Full dose anticoagulation.
* Known DPD-deficiency (special screening not required).
* Known glucuronidation-deficiency (special screening not required).
* Medical history of other malignant disease within 5 years prior to study entry, except for basalioma, and in-situ cervical carcinoma if treated with curative intent.
* Known alcohol or drug abuse.
* Medical or psychiatric condition which contradicts participation of study.
* Limited legal capacity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2007-01; Primary Completion 2014-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | approximate 6 months after randomisation

SECONDARY OUTCOMES:
Median progression free survival | approximate 6 months after randomisation
Median overall survival | approximate 3 years after randomisation
Secondary resection rate with curative intent | up to 3 months after end of treatment
Safety and toxicity (according to NCI-CTCAE) | approximate 6 months after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, MD, Principal Investigator — University of Munich - Klinikum Grosshadern
Locations (1):
- University of Munich - Klinikum Grosshadern, Munich, Germany

REFERENCES:
- [Derived] Stahler A, Modest DP, Stintzing S, Borelli B, Keller T, Held S, Fischer von Weikersthal L, Muller L, Graeven U, Decker T, Heintges T, Kahl C, Hoppe B, Kiani A, Kaiser F, Schwaner I, Fruehauf S, Karthaus M, Trarbach T, Klauschen F, Horst D, Cremolini C, Heinemann V. Individual Patient Data Meta-Analysis of Consensus Molecular Subtypes as Biomarkers of First-Line Treatment in RAS Wild-Type Metastatic Colorectal Cancer. J Clin Oncol. 2026 Jan;44(1):31-41. doi: 10.1200/JCO-25-00596. Epub 2025 Nov 18. PMID 41252656
- [Derived] Fischer LE, Stintzing S, von Weikersthal LF, Modest DP, Decker T, Kiani A, Kaiser F, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Giessen-Jung C, Uhlig J, Peuser B, Denzlinger C, Stahler A, Weiss L, Heinrich K, Held S, Jung A, Kirchner T, Heinemann V. Efficacy of FOLFIRI plus cetuximab vs FOLFIRI plus bevacizumab in 1st-line treatment of older patients with RAS wild-type metastatic colorectal cancer: an analysis of the randomised trial FIRE-3. Br J Cancer. 2022 Sep;127(5):836-843. doi: 10.1038/s41416-022-01854-y. Epub 2022 May 30. PMID 35637412
- [Derived] Heinemann V, von Weikersthal LF, Decker T, Kiani A, Kaiser F, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Moehler M, Scheithauer W, Held S, Miller-Phillips L, Modest DP, Jung A, Kirchner T, Stintzing S. FOLFIRI plus cetuximab or bevacizumab for advanced colorectal cancer: final survival and per-protocol analysis of FIRE-3, a randomised clinical trial. Br J Cancer. 2021 Feb;124(3):587-594. doi: 10.1038/s41416-020-01140-9. Epub 2020 Nov 6. PMID 33154570
- [Derived] Froelich MF, Petersen EL, Heinemann V, Norenberg D, Hesse N, Gesenhues AB, Modest DP, Sommer WH, Hofmann FO, Stintzing S, Holch JW. Impact of Size and Location of Metastases on Early Tumor Shrinkage and Depth of Response in Patients With Metastatic Colorectal Cancer: Subgroup Findings of the Randomized, Open-Label Phase 3 Trial FIRE-3/AIO KRK-0306. Clin Colorectal Cancer. 2020 Dec;19(4):291-300.e5. doi: 10.1016/j.clcc.2020.06.005. Epub 2020 Jun 22. PMID 32917529
- [Derived] Stintzing S, Wirapati P, Lenz HJ, Neureiter D, Fischer von Weikersthal L, Decker T, Kiani A, Kaiser F, Al-Batran S, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Moehler M, Scheithauer W, Held S, Modest DP, Jung A, Kirchner T, Aderka D, Tejpar S, Heinemann V. Consensus molecular subgroups (CMS) of colorectal cancer (CRC) and first-line efficacy of FOLFIRI plus cetuximab or bevacizumab in the FIRE3 (AIO KRK-0306) trial. Ann Oncol. 2019 Nov 1;30(11):1796-1803. doi: 10.1093/annonc/mdz387. PMID 31868905
- [Derived] Tokunaga R, Cao S, Naseem M, Lo JH, Battaglin F, Puccini A, Berger MD, Soni S, Millstein J, Zhang W, Stintzing S, Loupakis F, Cremolini C, Heinemann V, Falcone A, Lenz HJ. Prognostic Effect of Adenosine-related Genetic Variants in Metastatic Colorectal Cancer Treated With Bevacizumab-based Chemotherapy. Clin Colorectal Cancer. 2019 Mar;18(1):e8-e19. doi: 10.1016/j.clcc.2018.09.003. Epub 2018 Sep 13. PMID 30293873
- [Derived] Modest DP, Denecke T, Pratschke J, Ricard I, Lang H, Bemelmans M, Becker T, Rentsch M, Seehofer D, Bruns CJ, Gebauer B, Modest HI, Held S, Folprecht G, Heinemann V, Neumann UP. Surgical treatment options following chemotherapy plus cetuximab or bevacizumab in metastatic colorectal cancer-central evaluation of FIRE-3. Eur J Cancer. 2018 Jan;88:77-86. doi: 10.1016/j.ejca.2017.10.028. Epub 2017 Nov 28. PMID 29195117
- [Derived] Tejpar S, Stintzing S, Ciardiello F, Tabernero J, Van Cutsem E, Beier F, Esser R, Lenz HJ, Heinemann V. Prognostic and Predictive Relevance of Primary Tumor Location in Patients With RAS Wild-Type Metastatic Colorectal Cancer: Retrospective Analyses of the CRYSTAL and FIRE-3 Trials. JAMA Oncol. 2017 Feb 1;3(2):194-201. doi: 10.1001/jamaoncol.2016.3797. PMID 27722750
- [Derived] Stintzing S, Modest DP, Rossius L, Lerch MM, von Weikersthal LF, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Held S, Giessen-Jung C, Moehler M, Jagenburg A, Kirchner T, Jung A, Heinemann V; FIRE-3 investigators. FOLFIRI plus cetuximab versus FOLFIRI plus bevacizumab for metastatic colorectal cancer (FIRE-3): a post-hoc analysis of tumour dynamics in the final RAS wild-type subgroup of this randomised open-label phase 3 trial. Lancet Oncol. 2016 Oct;17(10):1426-1434. doi: 10.1016/S1470-2045(16)30269-8. Epub 2016 Aug 27. PMID 27575024
- [Derived] Michl M, Stintzing S, Fischer von Weikersthal L, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmueller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Hielscher J, Scholz M, Mueller S, Lerch MM, Modest DP, Kirchner T, Jung A, Heinemann V; FIRE-3 Study Group. CEA response is associated with tumor response and survival in patients with KRAS exon 2 wild-type and extended RAS wild-type metastatic colorectal cancer receiving first-line FOLFIRI plus cetuximab or bevacizumab (FIRE-3 trial). Ann Oncol. 2016 Aug;27(8):1565-72. doi: 10.1093/annonc/mdw222. Epub 2016 May 27. PMID 27234640
- [Derived] Modest DP, Stintzing S, von Weikersthal LF, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Held S, Mohler M, Jung A, Kirchner T, Heinemann V. Impact of Subsequent Therapies on Outcome of the FIRE-3/AIO KRK0306 Trial: First-Line Therapy With FOLFIRI Plus Cetuximab or Bevacizumab in Patients With KRAS Wild-Type Tumors in Metastatic Colorectal Cancer. J Clin Oncol. 2015 Nov 10;33(32):3718-26. doi: 10.1200/JCO.2015.61.2887. Epub 2015 Aug 10. PMID 26261259
- [Derived] Heinemann V, von Weikersthal LF, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Hielscher J, Scholz M, Muller S, Link H, Niederle N, Rost A, Hoffkes HG, Moehler M, Lindig RU, Modest DP, Rossius L, Kirchner T, Jung A, Stintzing S. FOLFIRI plus cetuximab versus FOLFIRI plus bevacizumab as first-line treatment for patients with metastatic colorectal cancer (FIRE-3): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Sep;15(10):1065-75. doi: 10.1016/S1470-2045(14)70330-4. Epub 2014 Jul 31. PMID 25088940